### UNIVERSITY OF CALIFORNIA LOS ANGELES STUDY INFORMATION SHEET

### Randomized Control Trial of Online Mental Health Promotion Program for University Students

Leslie Rith-Najarian, M.A. and Denise Chavira, Ph.D. from the Psychology Department and Elizabeth Gong-Guy, Ph.D., from Campus and Student Resilience at University of California, Los Angeles (UCLA) are conducting a research study.

You were invited as a possible participant in this study because you are currently 1) a student of the University of California, Los Angeles, 2) interested in the 8-week StriveWeekly programming, and 3) you are 18 years or older. Your participation in this research study is voluntary.

### Why is this study being done?

We are interested in learning more about how our program relates to student's mood, stress, and other cognitive and psychological experiences.

## What will happen if I participate in this research study? And what is the time required?

- You will complete an entry survey online by October 8, 2017 (approximately 8 minutes)
- You will be randomly assigned to access the 8-week online program in either Fall or Winter Quarter
- You will complete: program account creation, verification, and set-up (approximately 10 minutes)
- The activities and check-ins that you log on your online account will be included as part of our data collection
- You will complete a follow-up survey online in December (approximately 8 minutes)
- You will complete a follow-up survey online in March (approximately 8 minutes)

The questions in these surveys will ask about reasons for signing up, your psychological experiences, your motivation, and interaction with campus resources/services. In addition, survey data will be linked to data obtained from the UCLA Student Affairs Information and Research Office (SAIRO) using your student ID number (see further details under the confidentiality section below). All activities will be complete online and on a voluntary basis.

Are there any potential risks or discomforts that I can expect from this study? There are no anticipated risks or discomforts.

## Are there any potential benefits if I participate?

Based on prior research, students who complete the program may experience improvements in their anxiety or mood. In terms of benefits to society, the results of the research may advance our knowledge about disseminating effective healthy lifestyle programing on university campuses.

## Will I be paid for participating?

There is no direct payment for completing the surveys. However, your participation will earn your eligibility to be entered into the research study prize drawings

#### What is the prize drawing procedure?

Everyone who completes the entry and fall follow-up surveys be entered to win one of the research study prizes. The prizes will be one \$100 Amazon.com gift card and ten \$10 Amazon.com gift cards. A random number generator will be used to select the winners after the fall follow-up has closed. For the winter

follow-up survey, all participants will be entered into all 11 drawings for another set of Amazon.com gift cards with the same values.

Additional prizes will be offered as part of the program participation, in addition to the research survey prize drawing. All research study participants will have access to earn entry into those additional prize drawings by interacting with the program on a weekly basis during the quarter to which they are assigned (Fall or Winter). A random number generator will be used to select winners from the pool of eligible participants, according to these requirements:

-Weekly Prizes: are randomly given out weekly to 1-2 students. Who is entered into prize drawing: everyone who logs at least one activity that week and completes the Weekly Check-In (see the "Progress" tab on your dashboard) by Sunday at midnight of the respective week. -Finalist Prizes: 3-4 students will win gift cards or items of \$100-value. Who is entered into prize drawing: everyone who logs at least one activity every week and completes the follow-up survey. Once our [3 or 4] winners are drawn, they will get priority of prize choice based on total number of logged activities

-Finalist Reward Package: A packet of coupons and discount codes for local and online businesses. Who earns the prize: everyone who logs at least one activity every week.

What if I decline to participant in the research? Participation in the study is not required in order to participate in the raffle. If you would like to be entered into the drawing without participating in this study, you can contact Leslie at leslierrn@ucla.edu and you will be included within a single prize drawing for one of the \$10 Amazon.com gift cards.

Approximate odds of winning:

- For research participants: Best expected odds are 1:38 if the expected 420 students complete all surveys, and lowest expected odds are 1:76 if all students of the intended recruitment of 840 students complete both surveys.
  - Odds of weekly and finalist prizes are unpredictable as we do not know how many students will participate each week, but based on completion rates from prior studies, we expect odds to be 1:26 for winning a finalist prize and 1:12 for winning one of the weekly prizes if you complete all program weeks. If you complete all program weeks, you are guaranteed a Final Reward Package prize.
- For non-research participants entering the raffle: Highest expected odds are 1:420 if the expected 420 students complete all surveys, and lowest expected odds are 1:840 if all students of the intended recruitment of 840 students complete both surveys.

Selected prize winners will be contacted via email by Leslie Rith-Najarian (Principal Investigator).

## Will information about me and my participation be kept confidential?

Any information that is obtained in connection with this study and that can identify you will remain confidential. It will be disclosed only with your permission or as required by law. Confidentiality will be maintained for survey data using a secured database that is password protected. In addition, the online program's database is accessible only by the PI through a password protected account. The online platform uses a SSL certificate and has strong encryption for data transmit covering client to server communication and server to database communication.

The research team may not be able to keep confidential any disclosure or endorsement of thoughts to harm yourself. In the event that you indicate that you are thinking about killing yourself or you answer yes to a question about having thoughts about suicide, the research staff will ask you more questions about the thoughts. Depending on how intense your thoughts are or

how much you feel like hurting yourself, the research staff may provide you with referrals for treatment, work with you to contact your personal physician, trusted family member, or therapist to discuss your thoughts of harming yourself; or work with you on a plan that may include getting you to a hospital for safety.

Use of email address and student ID #: This information will be accessible only to authorized members of the research study team. Your email address will be used to connect your survey responses across questionnaires. Your student ID # will be used to connect your responses to your demographic information (gender, age, race/ethnicity, enrollment). The researchers of this study will not have access to your student records or other past survey responses. Instead, the demographic data will automatically be populated into our database through an agreement with Student Affairs Information and Research Office (SAIRO). Your responses to this survey will not be provided to SAIRO and will not be associated with your student record.

# What are my rights if I take part in this study?

- Your participation in this study is completely voluntary
- You can choose whether or not you want to be in this study, and you may withdraw your consent and discontinue participation at any time.
- Whatever decision you make, there will be no penalty to you, and no loss of benefits to which you were otherwise entitled.
- You may refuse to answer any questions that you do not want to answer and still remain in the study.

### Who can I contact if I have questions about this study?

#### The research team:

If you have any questions, comments or concerns about the research, you can talk to the one of the researchers.

Primary contact: Leslie Rith-Najarian – <u>leslierrn@ucla.edu</u> Faculty sponsor: Denise Chavira – dchavira@psych.ucla.edu

## UCLA Office of the Human Research Protection Program (OHRPP):

If you have questions about your rights as a research subject, or you have concerns or suggestions and you want to talk to someone other than the researchers, you may contact the UCLA OHRPP

- o by phone: (310) 206-2040;
- o by email: participants@research.ucla.edu
- o or by mail: Box 951406, Los Angeles, CA 90095-1406.